CLINICAL TRIAL: NCT02309216
Title: Whole-Body MRI in Suspected Victims of Abusive Head Trauma
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Susan Wootton, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0715
Record Dates: First submitted 2014-12-01; First posted 2014-12-05 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Shaken Baby Syndrome
MeSH Terms: conditions — Shaken Baby Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Whol-Body MRI scan

SUMMARY:
The purpose: to pilot whole-body MRI scanning in infants who are already getting brain MRI for suspected child abuse

Research design: prospective, blinded reading of Whole-Body MRI (WB-MRI) images during the routine care of the hospitalized infant with comparison to routine radiographic skeletal survey images

Procedures to be used: whole-body MRI images

Risks and potential benefits: no additional risk (the infant will be receiving and MRI of their brain as part of routine care, the additional images will be obtained at the same time without additional sedation); benefits to the infant include the identification of injuries which would have otherwise been missed by routine care importance of knowledge that may reasonably be expected to result: results from this study will potentially influence the use of radiographic skeletal survey and decrease the radiation exposure to infants being evaluated for suspected child abuse.

ELIGIBILITY:
Inclusion Criteria:

* younger than 12 months
* admitted to the hospital
* getting an MRI for suspected abusive head trauma

Exclusion Criteria:

-

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant inpatients being evaluated for suspected abusive head trauma who are already getting an MRI of the head and cervical spine.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
MRI findings of skeletal injuries, soft tissue injuries or visceral injuries | During hospitalization; MRI will typically be obtained on hospitalization day #2
  Whole Body MRI images will be read by a masked pediatric radiologist and compared with findings obtained by routine imaging and clinical evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States